CLINICAL TRIAL: NCT06209580
Title: Phase I/II Study of AMT-253 in Patients With Unresectable or Metastatic Malignant Melanoma and Other Advanced Solid Tumors
Brief Title: AMT-253 in Patients With Advanced Solid Tumours
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Multitude Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMT-253-02
Record Dates: First submitted 2024-01-08; First posted 2024-01-17 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Malignant Melanoma; Advanced Solid Tumors
MeSH Terms: conditions — Melanoma | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): AMT-253 Dose Escalation
  Interventions: Drug: AMT-253 for injection
- Arm 2 (Experimental): AMT-253 Dose Expansion
  Interventions: Drug: AMT-253 for injection

INTERVENTIONS:
Drug: AMT-253 for injection — Administered intravenously

SUMMARY:
This is a non-randomized, open-label, multicenter Phase I/II study of AMT-253 in patients with Unresectable or Metastatic Malignant Melanoma and other Advanced Solid Tumors. This study include phase I dose escalation and phase II dose expansion.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients must be willing and able to understand and sign the ICF, and to adhere to the study visit schedule and other protocol requirements.
* 2. Patients with histologically confirmed melanoma or other advanced solid tumor.
* 3. Patients who have undergone at least one systemic therapy and have radiologically or clinically determined progressive disease (PD) during or after most recent line of therapy, and for whom no further standard therapy is available, or who are intolerable to standard therapy.
* 4. Patients must have at least one measurable lesion as per RECIST version 1.1.
* 5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* 6. Life expectancy ≥ 3 months.
* 7. Patients must have adequate organ function
* 8. Women of child bearing potential (WCBP), defined as a sexually mature woman who has not undergone surgical sterilization or who has not been naturally postmenopausal for at least 12 consecutive months must agree to use two effective contraceptive methods while on study treatment and for at least twelve weeks after the last dose of the IMP.
* 9. WCBP must have a negative serum pregnancy test within 7 days prior to first dose of the IMP.
* 10. Male patients must agree to use a latex condom, even if they had a successful vasectomy, while on study treatment and for at least twelve weeks after the last dose of the IMP.
* 11. Male patients must agree not to donate sperm, and female patients must agree not to donate eggs, while on study treatment and for at least 12 weeks after the last dose of the IMP.
* 12. Availability of tumor tissue sample at screening.

Exclusion Criteria:

* 1. Prior treatment with any agent that has the same target.
* 2. Central nervous system (CNS) metastasis.
* 3. Active or chronic skin disorder requiring systemic therapy.
* 4. History of Steven's Johnson's syndrome or toxic epidermal necrolysis syndrome.
* 5. Persistent toxicities from previous systemic anti-neoplastic treatments of Grade >1.
* 6. Systemic anti-neoplastic therapy within five half-lives or 21 days, whichever is shorter, prior to first dose of the IMP.
* 7. Major surgery within 28 days prior to first dose of the IMP, or no recovery from side effects of such intervention.
* 8. Significant cardiac disease, such as recent myocardial infarction or acute coronary syndromes, congestive heart failure， uncontrolled hypertension, uncontrolled cardiac arrhythmias.
* 9. History of thromboembolic or cerebrovascular events, including transient ischemic attacks, cerebrovascular accidents, deep vein thrombosis, or pulmonary emboli within six months prior to first dose of the IMP.
* 10. Acute and/or clinically significant bacterial, fungal or viral infection including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus (HIV).
* 11. Administration of a live vaccine within 28 days prior to the administration of the first dose of the IMP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
DLTs | 21 days after first dose
  Incidence of dose limiting toxicities
AEs | Up to 24 months
  Type, incidence and severity of Adverse Events
SAEs | Up to 24 months
  Type, incidence and severity Serious Adverse Events (SAEs)
ORR | Up to 24 months
  Overall response rate assessed by the investigator according to RECIST version 1.1

SECONDARY OUTCOMES:
Cmax | Up to 24 months
  aximum concentration (Cmax)
Tmax | Up to 24 months
  time to peak drug concentration
AUC | Up to 24 months
  Area Under the Curve
t1/2 | Up to 24 months
  terminal half-life of the ADC, total antibody and free payload
ADAs | Up to 24 months
  Specification and quantification of anti-drug antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China